CLINICAL TRIAL: NCT05327816
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2a Study for Safety and Immunogenicity Evaluations of Various RSV.preF-based Vaccine Formulations in Adults Aged 60 Years and Older
Brief Title: A Study of Various Respiratory Syncytial Virus (RSV) Pre-Fusion (preF)-Based Vaccine Formulations in Adults Aged 60 Years and Older
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on recent study data from VAC18193, it was decided to terminate the study. There are no underlying safety concerns to terminate VAC18195RSV1001
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109184; VAC18195RSV1001 (Other: Janssen Vaccines & Prevention B.V.); 2022-001015-14 (EudraCT Number)
Record Dates: First submitted 2022-04-13; First posted 2022-04-14 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus-associated Lower Respiratory Tract Disease Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Arm 1a: Respiratory Syncytial Virus (RSV) preFusion (preF) Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in cohort (C) 1 (Group [G] 1) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 1b: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 1-4) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 1c: Placebo (Experimental): Participants will receive single dose of placebo in C 1 (G 1-4) and C 2 through intramuscular injection on Day 1.
  Interventions: Drug: Placebo
- Arm 2: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 2) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 3: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 2) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 4: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 2) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 5: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 2) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 6: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 2) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 7: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 3) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 8: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 3) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 9: RSV preF Based Vaccine (Experimental): Participants will receive single dose of mixture of RSV preF-based vaccine in C 1 (G 4) and C 2 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 10: RSV preF Based Vaccine (Experimental): Participants will receive a single dose of selected formulation (based on C 1 and 2 results) in C 3 through intramuscular injection on Day 1.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 11a: RSV preF Based Vaccine and Placebo (Experimental): Participants in C 3 will receive a single dose of first vaccination with selected formulation (as per data C1 and 2) plus placebo on Day 1 and re-vaccination with selected formulation whenever revaccination would be needed through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine; Drug: Placebo
- Arm 11b: RSV preF Based Vaccine and Placebo (Experimental): Participants in C 3 will receive a single dose of first vaccination with selected formulation (as per data from C 1 and 2) plus placebo on Day 1 and re-vaccination with placebo whenever revaccination would be needed through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine; Drug: Placebo
- Arm 12: RSV preF Based Vaccine and Placebo (Experimental): Participants in C 3 will receive first vaccination with placebo on Day 1 and re-vaccination with selected formulation (as per data from C 1 and 2) whenever revaccination would be needed through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine; Drug: Placebo
- Arm 13: RSV preF Based Vaccine (Experimental): Participants in C 3 will receive the mixture of RSV preF-based vaccine plus placebo on Day 1 through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine; Drug: Placebo
- Arm 14: RSV preF Based Vaccine (Experimental): Participants in C 4 will receive first vaccination with selected formulation (as per data from C 1 and 2) on Day 1 and re-vaccination with selected formulation whenever revaccination would be needed through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine
- Arm 15: RSV preF Based Vaccine and Placebo (Experimental): Participants in C 4 will receive first vaccination with selected formulation (as per data from C 1 and 2) on Day 1 and re-vaccination with placebo whenever revaccination would be needed through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine; Drug: Placebo
- Arm 16: RSV preF Based Vaccine and Placebo (Experimental): Participants in C 4 will receive first vaccination with placebo on Day 1 and re-vaccination with selected formulation (as per data from C 1 and 2) whenever revaccination would be needed through intramuscular injection.
  Interventions: Biological: RSV preF-based Vaccine; Drug: Placebo

INTERVENTIONS:
Biological: RSV preF-based Vaccine — RSV preF-based vaccine will be administered as intramuscular injection.
  Arms: Arm 10: RSV preF Based Vaccine; Arm 11a: RSV preF Based Vaccine and Placebo; Arm 11b: RSV preF Based Vaccine and Placebo; Arm 12: RSV preF Based Vaccine and Placebo; Arm 13: RSV preF Based Vaccine; Arm 14: RSV preF Based Vaccine; Arm 15: RSV preF Based Vaccine and Placebo; Arm 16: RSV preF Based Vaccine and Placebo; Arm 1a: Respiratory Syncytial Virus (RSV) preFusion (preF) Based Vaccine; Arm 1b: RSV preF Based Vaccine; Arm 2: RSV preF Based Vaccine; Arm 3: RSV preF Based Vaccine; Arm 4: RSV preF Based Vaccine; Arm 5: RSV preF Based Vaccine; Arm 6: RSV preF Based Vaccine; Arm 7: RSV preF Based Vaccine; Arm 8: RSV preF Based Vaccine; Arm 9: RSV preF Based Vaccine
Drug: Placebo — Placebo will be administered as intramuscular injection.
  Arms: Arm 11a: RSV preF Based Vaccine and Placebo; Arm 11b: RSV preF Based Vaccine and Placebo; Arm 12: RSV preF Based Vaccine and Placebo; Arm 13: RSV preF Based Vaccine; Arm 15: RSV preF Based Vaccine and Placebo; Arm 16: RSV preF Based Vaccine and Placebo; Arm 1c: Placebo

SUMMARY:
The purpose of the study is to evaluate safety and immunogenicity of various respiratory syncytial virus (RSV) pre-Fusion (preF)-based vaccine components followed by expanded safety evaluation and durability/revaccination evaluation of the selected RSV preF-based vaccine formulation in participants aged greater than or equal to (>=) 60 years in stable health.

DETAILED DESCRIPTION:
RSV is an important cause of serious respiratory infections in adults aged 60 years and older. The current study is divided into four cohorts, evaluating various doses and combinations of RSV preF-based vaccines. Cohort 1 will assess the safety and reactogenicity of different RSV preF-based vaccines. Cohort 2 is an expansion of cohort 1 and will assess both safety and immunogenicity of these different RSV vaccines. based on C1 and 2 data the optimal vaccine composition will be selected and further evaluated in Cohort 3 and 4 including durability and revaccination. Cohort 3 will accumulate safety data on the selected vaccine and optimize its formulation. Cohort 4 is an expansion of several arms in cohort 3, aimed to understand the durability of the immune response induced by the selected vaccine, and to explore the possibility for revaccination.

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's clinical judgment, participant must be in stable health at the time of vaccination. Participants may have underlying illnesses such as hypertension, congestive heart failure, chronic obstructive pulmonary disease (COPD), Type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are stable at the time of vaccination, and these conditions receive routine follow-up by the participant's healthcare provider.
* Participants will be included on the basis of physical examination, medical history, and vital signs performed between informed consent form (ICF) signature and vaccination
* For participants in Cohorts 1 and 2 only: Participant must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the laboratory screening tests are outside the laboratory normal reference ranges and additionally within the limits of toxicity Grade 2 according to the United States Food and Drug Administration (US FDA) toxicity tables (that is, for tests in the FDA table), the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Agrees not to donate blood from the time of vaccination through 3 months after vaccination
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* History of malignancy within 5 years before screening not in the following categories: a) Participants with squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix may be enrolled at the discretion of the investigator; b) Participants with a history of malignancy within 5 years before screening, with minimal risk of recurrence per investigator's judgment, can be enrolled
* Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine components
* Per medical history, participant has chronic active hepatitis B or hepatitis C infection, human immunodeficiency viruses (HIV) type 1 or type 2 infection, acute polyneuropathy (example, Guillain-Barré syndrome) or chronic idiopathic demyelinating polyneuropathy
* Participant is in receipt of, or planning to receive, licensed live attenuated vaccine within 28 days before and after study vaccinations; other licensed vaccines (that is, not live such as, influenza, tetanus, hepatitis A or B, rabies) within 14 days before and after study vaccinations
* Received treatment with immunoglobulins expected to impact the vaccine-induced immune response (including monoclonal antibodies [MAbs] for chronic underlying conditions) in the 2 months; immunoglobulins specific to respiratory syncytial virus (RSV), human metapneumovirus, or parainfluenza viruses in the 12 months; apheresis therapies in the 4 months; or blood products in the 4 months prior to study vaccination or has any plans to receive such treatment during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (11):
- United States (11):
  - Ark Clinical Research, Long Beach, California
  - Accel Research Sites, DeLand, Florida
  - Floridian Clinical Research LLC, Miami Lakes, Florida
  - Heartland Research Associates, an AMR Company, Wichita, Kansas
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - The Center for Pharmaceutical Research (CPR), Kansas City, Missouri
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee
  - Tekton Research Inc., Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated on sponsor's decision, hence, participants were enrolled in Cohort 1 only. Cohorts 2, 3, and 4 were not initiated. Participants enrolled in Cohort 1 completed visit up to Day 183 (6-months post vaccination) and safety evaluations were performed only for Cohort 1. Since the study was terminated prior to Cohort 2 enrolment and the data was planned for combined Cohorts 1 and 2, samples collected in Cohort 1 alone were not tested and no immunogenicity testing was performed.
Groups:
- Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg: Participants received single intramuscular (IM) injections of adenovirus serotype 26 respiratory syncytial virus-B prefusion-F2 protein (Ad26.RSV-B.preF2) 1*10^11 viral particles (vp) and RSV-B.preF protein 150 micrograms (mcg) on Day 1.
- Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg: Participants received single IM injections of adenovirus serotype 26 respiratory syncytial virus-A prefusion-F protein (Ad26.RSV-A.preF) 1*10^11 vp and RSV-A.preF protein 150 mcg on Day 1.
- Arm 1c (Cohort 1): Pooled Placebo: Participants received a single IM injection of placebo on Day 1.
- Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg: Participants received single IM injections of RSV-A.preF protein 150 mcg and RSV-B.preF protein 150 mcg on Day 1.
- Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg: Participants received single IM injections of Ad26.RSV-A.preF 2.5*10^10 vp, Ad26.RSV-B.preF2 2.5 *10^10 vp, RSV-A.preF protein 150 mcg, and RSV-B.preF protein 150 mcg on Day 1.
- Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg: Participants received single IM injections of Ad26.RSV-A.preF 5*10^10 vp, Ad26.RSV-B.preF2 5 *10^10 vp, RSV-A.preF protein 150 mcg, and RSV-B.preF protein 150 mcg on Day 1.
- Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg: Participants received single IM injections of Ad26.RSV-A.preF 1*10^11 vp and RSV-A.preF protein 300 mcg on Day 1.
- Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg: Participants received single IM injections of Ad26.RSV-A.preF 1*10^11 vp, RSV-A.preF protein 150 mcg, and RSV-B.preF protein 150 mcg on Day 1.
- Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg: Participants received single IM injections of Ad26.RSV-A.preF 1*10^11 vp, Ad26.RSV-B.preF2 5*10^10 vp, RSV-A.preF protein 150 mcg, and RSV-B.preF protein 150 mcg on Day 1.
- Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg: Participants received single IM injections of Ad26.RSV-A.preF 1.5*10^11 vp and RSV-A.preF protein 300 mcg on Day 1.
- Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg: Participants received single IM injections of Ad26.RSV-A.preF 1*10^11 vp, Ad26.RSV-B.preF2 1*10^11 vp, RSV-A.preF protein 150 mcg, and RSV-B.preF protein 150 mcg on Day 1.
Period: Overall Study
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Treated (Full Analysis Set) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 11 | 12 | 12 | 12 | 11 | 11 | 11 | 11 | 11 | 11 | 12
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received the study vaccine, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (5.42) | 67.8 (5.01) | 66.2 (5.65) | 69.3 (3.39) | 65.7 (4.94) | 67.4 (4.83) | 68.5 (6.12) | 64.8 (4.14) | 66.3 (3.04) | 65.4 (4.4) | 65.5 (3.78) | 66.9 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 6 | 10 | 6 | 6 | 6 | 9 | 7 | 6 | 5 | 77
  Male | 3 | 5 | 6 | 2 | 6 | 6 | 5 | 2 | 4 | 6 | 7 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 7
  Not Hispanic or Latino | 12 | 11 | 11 | 12 | 12 | 12 | 11 | 9 | 11 | 11 | 10 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 1 | 2 | 1 | 1 | 3 | 3 | 1 | 2 | 2 | 18
  White | 12 | 10 | 11 | 10 | 10 | 10 | 8 | 8 | 10 | 10 | 10 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From Day 1 up to 6 months post vaccination (up to Day 183)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12
Participants | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Number of participants with AESIs were reported. Thrombosis with thrombocytopenia syndrome (TTS) were considered as potential AESIs.
Time Frame: From Day 1 up to 6 months post vaccination (up to Day 183)
Population: The FAS included all participants who received the study vaccine, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AEs)
Description: Number of participants with solicited local and systemic AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Solicited systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post vaccination (Day 8)
Population: The FAS included all participants who received the study vaccine, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12
Participants
  Solicited Local AEs | 6 | 8 | 5 | 7 | 8 | 10 | 7 | 8 | 9 | 11 | 7
  Solicited Systemic AEs | 9 | 8 | 7 | 8 | 9 | 10 | 7 | 10 | 10 | 10 | 7

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: Number of participants with unsolicited AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant were not specifically questioned in the participant diary.
Time Frame: 28 days post vaccination (Day 29)
Population: The FAS included all participants who received the study vaccine, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12 | 12
Participants | 5 | 2 | 4 | 3 | 4 | 0 | 2 | 1 | 4 | 5 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 up to 6 months post vaccination (up to Day 183)
Description: The full analysis set (FAS) included all participants who received the study vaccine, regardless of the occurrence of protocol deviations.
Arm/Group | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg | Arm 1c (Cohort 1): Pooled Placebo | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/11 | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12 | 1/12 | 0/12 | 0/12 | 1/11 | 1/11 | 1/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 9/12 | 10/12 | 10/12 | 10/12 | 11/12 | 8/11 | 11/11 | 10/11 | 11/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg (N=12) | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg (N=12) | Arm 1c (Cohort 1): Pooled Placebo (N=12) | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg (N=12) | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg (N=12) | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg (N=12) | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg (N=11) | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg (N=11) | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg (N=11) | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg (N=12) | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg (N=12)
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1a (Cohort 1): Ad26.RSV-B.PreF2 1*10^11 vp + RSV-B.PreF Protein 150 mcg (N=12) | Arm 1b (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 150 mcg (N=12) | Arm 1c (Cohort 1): Pooled Placebo (N=12) | Arm 2 (Cohort 1): RSV-A.PreF Protein 150 mcg + RSV-B.PreF Protein 150 mcg (N=12) | Arm 3 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 2.5*10^10 vp + RSV-A.PreF/RSV-B.PreF 150 mcg (N=12) | Arm 4 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 5*10^10 vp + RSV-A.PreF /RSV-B.PreF 150 mcg (N=12) | Arm 5 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF Protein 300 mcg (N=11) | Arm 6 (Cohort 1): Ad26.RSV-A.PreF 1*10^11 vp + RSV-A.PreF and RSV-B.PreF at 150 mcg (N=11) | Arm 7 (Cohort 1):Ad26.RSV-A.PreF 1*10^11vp/Ad26.RSV-B.preF2 5*10^10vp + RSV-A.Pre/RSV-B.PreF 150 mcg (N=11) | Arm 8 (Cohort 1): Ad26.RSV-A.PreF 1.5*10^11 vp +RSV-A.PreF Protein 300 mcg (N=12) | Arm 9 (Cohort 1): Ad26.RSV-A.PreF/Ad26.RSV-B.preF2 1*10^11 vp + RSV-A.PreF/RSV-B.PreF 150 mcg (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 3 | 4 | 3 | 4 | 3 | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1
Fatigue (General disorders) | 6 | 7 | 6 | 5 | 7 | 8 | 5 | 9 | 8 | 10 | 7
Injection Site Bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 2 | 1 | 3 | 2 | 1 | 5 | 3 | 2
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Tenderness (General disorders) | 6 | 8 | 5 | 7 | 8 | 10 | 7 | 8 | 9 | 11 | 7
Covid-19 (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea Pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil Count Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 4 | 6 | 8 | 8 | 6 | 9 | 8 | 9 | 6
Headache (Nervous system disorders) | 5 | 6 | 5 | 3 | 4 | 4 | 6 | 8 | 8 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated on sponsor's decision, hence, participants were enrolled in Cohort 1 only. Cohorts 2, 3, and 4 were not initiated. Participants enrolled in Cohort 1 completed visit up to Day 183 (6-months post vaccination) and safety evaluations were performed only for Cohort 1. Since the study was terminated prior to Cohort 2 enrolment and the data was planned for combined Cohorts 1 and 2, samples collected in Cohort 1 alone were not tested and no immunogenicity testing was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT05327816/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT05327816/SAP_001.pdf